CLINICAL TRIAL: NCT04309123
Title: Pilot Study of TransAeris® System in Surgical Patients at Risk of Prolonged Mechanical Ventilation
Acronym: TRANSITION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Synapse Biomedical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-1000-100
Record Dates: First submitted 2020-03-12; First posted 2020-03-16 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Ventilator-Induced Diaphragm Dysfunction
Keywords: VIDD

STUDY DESIGN:
Intervention Model Description: Open label observational study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment (Experimental): TransAeris stimulation therapy adjunctive to continued mechanical ventilation will begin 24 hours after leaving the operating room, if subject remains on mechanical ventilation. TransAeris stimulator settings (stimulus intensity, stimulus frequency, and burst on/off) will be programmed to optimize diaphragm recruitment without compromising patient comfort.
  Interventions: Device: TransAeris System

INTERVENTIONS:
Device: TransAeris System — The TransAeris System is a temporary percutaneous intramuscular diaphragm stimulator intended for patients at risk of or on prolonged positive pressure mechanical ventilation. TransAeris is indicated for use in the prevention and treatment of ventilator-induced diaphragm dysfunction (VIDD).

SUMMARY:
This study will be conducted as a pilot trial of the TransAeris system for the prevention and treatment of ventilator-induced diaphragm dysfunction (VIDD) in patients identified prior to surgery to be at greater risk of prolonged mechanical ventilation (PMV).

DETAILED DESCRIPTION:
This pilot study is an open label observational study in adult open cardiac surgery patients. Eligible patients from whom informed consent is obtained and electrodes are successfully implanted are enrolled in the study. All subjects will be implanted with the TransLoc electrodes during their primary surgery. Following admission to the ICU, diaphragm EMG recording will begin and continue until TransAeris use begins or until discharge from the ICU. TransAeris stimulation therapy adjunctive to continued MV will begin 24 hours after leaving the operating room. TransAeris stimulator settings (stimulus intensity, stimulus frequency, and burst on/off) will be programmed to optimize diaphragm recruitment without compromising patient comfort.

When deemed ready by the physician, the subject will perform a spontaneous breathing trial (SBT). Diaphragm EMG will be recorded for the first 15 minutes of an SBT, when performed with study staff available, then TransAeris therapy will continue. If an SBT is not performed on a day or performed when study staff is not available, a diaphragm EMG will be recorded for 15 minutes and then TransAeris therapy will be resumed. If the subject fails the SBT or the physician determines the subject is inappropriate for extubation, TransAeris stimulation therapy will continue. Prior to leaving the ICU, diaphragm EMG will be recorded for 15 minutes and the TransLoc electrodes will be removed. Subjects that reach Day 30 after implantation will stop TransAeris therapy. Diaphragm EMG will be recorded for 15 minutes and the TransLoc electrodes will be removed prior to the end of Day 30.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is undergoing an open cardiac procedure by median sternotomy
2. Subject is at risk of prolonged mechanical ventilation ≥ 24H
3. Subject is at least 22 years of age
4. Informed consent has been obtained from the subject or designated representative

Exclusion Criteria:

1. Subject is on invasive mechanical ventilation prior to procedure
2. Subject has known or pre-existing phrenic nerve paralysis
3. Subject has progressive, non-reversible neuromuscular disease affecting the diaphragm
4. Subject is pregnant or lactating
5. Subject is actively participating in another clinical study which could affect outcomes in this study

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 60 Days
  Incidence of Serious Device Related Adverse Events

SECONDARY OUTCOMES:
Duration on Mechanical Ventilation | 30 Days
  Time on Mechanical Ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Raymond P Onders, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No